CLINICAL TRIAL: NCT01980017
Title: A Prospective Cluster-Randomized Trial to Implement the Ottawa Model for Smoking Cessation in Diabetes Education Programs.
Brief Title: Evaluation of the Ottawa Model for Smoking Cessation in Diabetes Education Programs
Acronym: OMSCinDEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20130177-01H
Record Dates: First submitted 2013-11-01; First posted 2013-11-08 (Estimated); Results first posted 2022-04-20 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Pre-diabetic; Diabetic Type II Mellitus
Keywords: Diabetes Type 2 Mellitus; Ottawa Model for Smoking Cessation; Diabetes Education Programs
MeSH Terms: conditions — Glucose Intolerance; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Wait-Listed Control Group (No Intervention): Usual care for smoking cessation
- Ottawa Model for Smoking Cessation (Experimental): Ottawa Model for Smoking Cessation
  Interventions: Behavioral: Ottawa Model for Smoking Cessation

INTERVENTIONS:
Behavioral: Ottawa Model for Smoking Cessation
  Arms: Ottawa Model for Smoking Cessation

SUMMARY:
The incidence of type 2 diabetes mellitus (T2DM) is increasing rapidly. The combination of T2DM and smoking is particularly lethal, as smokers with T2DM are significantly more likely to develop a number of health related complications. Community-based diabetes education programs (DEPs) have been developed to support patient self-care behaviours (e.g. adherence to oral medications, insulin therapy, nutrition management, regular blood glucose monitoring, and physical activity); however, specific assistance for smoking cessation is rarely provided. Our investigative team has developed a knowledge transfer and practice change process to introduce evidence-based interventions for smoking cessation into clinical practice settings. This process is known as the Ottawa Model for Smoking Cessation (OMSC). Investigators believe there is an opportunity to use the OMSC intervention to dramatically enhance the effectiveness of DEPs in addressing smoking cessation among smokers with T2DM, and in so doing, improve quit rates in this high risk population.

The purpose of this project is to evaluate the effectiveness of the Ottawa Model for Smoking Cessation (OMSC) intervention in multiple diabetes education programs (DEPs) in Ontario. A two-level recruitment strategy will be employed. Eighteen DEPs will be recruited, and then a consecutive sample of eligible smoker-patients will be recruited from each DEP over a 6-month recruitment period. Investigators want to test the impact of the OMSC intervention on quit rates among smokers with diabetes and pre-diabetes referred to these programs. Investigators will conduct a matched-pair cluster design trial at 18 DEPs in Ontario. These sites will be matched based on number of annual referrals for diabetes education (≤ 500/year or > 500/year). Within each pair, sites will be allocated randomly to either OMSC intervention or control group. Following randomization, the OMSC program will be implemented at the intervention sites over a 6-month period. Following the implementation period, a consecutive sample of smokers will be recruited from both OMSC intervention and control DEPs over a 6-month recruitment period. It is estimated that this will yield a sample of approximately 445 smokers in each of the OMSC intervention and control groups. The primary outcome will be the biochemically-validated 7-day point prevalence abstinence rate six months after an index visit to the DEP. Secondary outcomes will include: rates of identification and intervention of smokers, and diabetes educators' attitudes, confidence, and perceptions of barriers and facilitators to implementing smoking cessation support as part of routine care.

If proven effective, the OMSC is appropriate for implementation in DEPs across Canada and could have profound impacts on patient and community health.

ELIGIBILITY:
Inclusion Criteria:

* The patient has been referred to DEP for T2DM diabetes or pre-diabetes.
* The patient is a current smoker (self-report of daily smoking a minimum of 1 cigarette per day in the 30 days preceding recruitment).
* The patient is aged between 18 years and 80 years.

Exclusion Criteria:

* The patient is currently involved in any other smoking cessation intervention.
* The patient is able to read and understand French or English.
* The patient is able to and willing to provide informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 313 (Actual)
Dates: Start 2013-07; Primary Completion 2016-10-18 (Actual); Study Completion 2017-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Reid, PhD., MBA, Principal Investigator — Ottawa Heart Institute Research Corporation; Andrew Pipe, MD, FRCPC, Study Chair — Ottawa Heart Institute Research Corporation; Oh Paul, MD, FRCPC, Study Chair — Toronto Rehabilitation Institute; Anil Gupta, MD, FRCPC, Study Chair — Trillium Heath Centre; Kocourek Jana, MA, Study Chair — Ottawa Heart Institute Research Corporation; Mullen Kerri-Anne, MSc., Study Chair — Ottawa Heart Institute Research Corporation; Aiken Debbie, BScN, Study Chair — Ottawa Heart Institute Research Corporation; Tulloch Heather, Ph.D., Psych., Study Chair — Ottawa Heart Institute Research Corporation; David Arbeau, BA, BTech, RT, Study Chair — Horizon Health Network; Malcolm Janine, MD, FRCPC, Study Chair — Faculty of Medicine, University of Ottawa
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada

REFERENCES:
- [Background] Willi C, Bodenmann P, Ghali WA, Faris PD, Cornuz J. Active smoking and the risk of type 2 diabetes: a systematic review and meta-analysis. JAMA. 2007 Dec 12;298(22):2654-64. doi: 10.1001/jama.298.22.2654. PMID 18073361
- [Background] Doll R, Peto R, Boreham J, Sutherland I. Mortality in relation to smoking: 50 years' observations on male British doctors. BMJ. 2004 Jun 26;328(7455):1519. doi: 10.1136/bmj.38142.554479.AE. Epub 2004 Jun 22. PMID 15213107
- [Background] Stamler J, Vaccaro O, Neaton JD, Wentworth D. Diabetes, other risk factors, and 12-yr cardiovascular mortality for men screened in the Multiple Risk Factor Intervention Trial. Diabetes Care. 1993 Feb;16(2):434-44. doi: 10.2337/diacare.16.2.434. PMID 8432214
- [Background] Grimshaw JM, Eccles MP, Lavis JN, Hill SJ, Squires JE. Knowledge translation of research findings. Implement Sci. 2012 May 31;7:50. doi: 10.1186/1748-5908-7-50. PMID 22651257
- [Background] Reid RD, Pipe AL, Quinlan B. Promoting smoking cessation during hospitalization for coronary artery disease. Can J Cardiol. 2006 Jul;22(9):775-80. doi: 10.1016/s0828-282x(06)70294-x. PMID 16835672
- [Background] Reid RD, Pipe AL, Quinlan B, Oda J. Interactive voice response telephony to promote smoking cessation in patients with heart disease: a pilot study. Patient Educ Couns. 2007 Jun;66(3):319-26. doi: 10.1016/j.pec.2007.01.005. Epub 2007 Mar 1. PMID 17336026
- [Background] Reid RD, Mullen KA, Slovinec D'Angelo ME, Aitken DA, Papadakis S, Haley PM, McLaughlin CA, Pipe AL. Smoking cessation for hospitalized smokers: an evaluation of the "Ottawa Model". Nicotine Tob Res. 2010 Jan;12(1):11-8. doi: 10.1093/ntr/ntp165. Epub 2009 Nov 10. PMID 19903737
- [Background] Reid RD, Mullen KA, Pipe AL. Systematic approaches to smoking cessation in the cardiac setting. Curr Opin Cardiol. 2011 Sep;26(5):443-8. doi: 10.1097/HCO.0b013e3283497499. PMID 21730824
- [Background] SRNT Subcommittee on Biochemical Verification. Biochemical verification of tobacco use and cessation. Nicotine Tob Res. 2002 May;4(2):149-59. doi: 10.1080/14622200210123581. No abstract available. PMID 12028847
- [Background] Donner A, Donald A. Analysis of data arising from a stratified design with the cluster as unit of randomization. Stat Med. 1987 Jan-Feb;6(1):43-52. doi: 10.1002/sim.4780060106. PMID 3576016
- [Background] Thompson SG, Pyke SD, Hardy RJ. The design and analysis of paired cluster randomized trials: an application of meta-analysis techniques. Stat Med. 1997 Sep 30;16(18):2063-79. doi: 10.1002/(sici)1097-0258(19970930)16:183.0.co;2-8. PMID 9308132
- [Background] Campbell MK, Mollison J, Grimshaw JM. Cluster trials in implementation research: estimation of intracluster correlation coefficients and sample size. Stat Med. 2001 Feb 15;20(3):391-9. doi: 10.1002/1097-0258(20010215)20:33.0.co;2-z. PMID 11180309
- [Background] Papadakis S, Aitken D, Gocan S, Riley D, Laplante MA, Bhatnagar-Bost A, Cousineau D, Simpson D, Edjoc R, Pipe AL, Sharma M, Reid RD. A randomised controlled pilot study of standardised counselling and cost-free pharmacotherapy for smoking cessation among stroke and TIA patients. BMJ Open. 2011 Nov 28;1(2):e000366. doi: 10.1136/bmjopen-2011-000366. Print 2011. PMID 22123923
- [Background] Reid RD, Pipe A, Dafoe WA. Is telephone counselling a useful addition to physician advice and nicotine replacement therapy in helping patients to stop smoking? A randomized controlled trial. CMAJ. 1999 Jun 1;160(11):1577-81. PMID 10373999
- [Background] Reid RD, Pipe AL. A telephone-based support program for over-the-counter nicotine patch users. Can J Public Health. 1999 Nov-Dec;90(6):397-8. doi: 10.1007/BF03404144. No abstract available. PMID 10680265
- [Background] Slovinec D'Angelo ME, Reid RD, Hotz S, Irvine J, Segal RJ, Blanchard CM, Pipe A. Is stress management training a useful addition to physician advice and nicotine replacement therapy during smoking cessation in women? Results of a randomized trial. Am J Health Promot. 2005 Nov-Dec;20(2):127-34. doi: 10.4278/0890-1171-20.2.127. PMID 16295704
- [Background] Rigotti NA, Pipe AL, Benowitz NL, Arteaga C, Garza D, Tonstad S. Efficacy and safety of varenicline for smoking cessation in patients with cardiovascular disease: a randomized trial. Circulation. 2010 Jan 19;121(2):221-9. doi: 10.1161/CIRCULATIONAHA.109.869008. Epub 2010 Jan 4. PMID 20048210
- [Background] Campbell MK, Piaggio G, Elbourne DR, Altman DG; CONSORT Group. Consort 2010 statement: extension to cluster randomised trials. BMJ. 2012 Sep 4;345:e5661. doi: 10.1136/bmj.e5661. No abstract available. PMID 22951546
- [Derived] Reid RD, Malcolm J, Wooding E, Geertsma A, Aitken D, Arbeau D, Blanchard C, Gagnier JA, Gupta A, Mullen KA, Oh P, Papadakis S, Tulloch H, LeBlanc AG, Wells GA, Pipe AL. Prospective, Cluster-Randomized Trial to Implement the Ottawa Model for Smoking Cessation in Diabetes Education Programs in Ontario, Canada. Diabetes Care. 2018 Mar;41(3):406-412. doi: 10.2337/dc17-1809. Epub 2017 Dec 21. PMID 29269509

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Wait-Listed Control Group | Ottawa Model for Smoking Cessation
Started | 114 | 199
Completed | 84 | 177
Not Completed | 30 | 22
Not completed — Lost to Follow-up | 30 | 21
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Wait-Listed Control Group | Ottawa Model for Smoking Cessation | Total
Number analyzed (Participants) | 114 | 199 | 313
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 76 | 136 | 212
  >=65 years | 38 | 63 | 101
Age, Continuous [Mean (Full Range); unit: years] | 54.9 [23 to 72] | 54 [22 to 78] | 54.4 [22 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 89 | 138
  Male | 65 | 110 | 175
Region of Enrollment [Number; unit: participants]
  Canada | 114 | 199 | 313

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Self Report of Not Smoking (Even a Puff) in the Last 7 Days + CO <10ppm
Description: The OMSC intervention will increase carbon monoxide (CO) validated 7-day point prevalence abstinence rates at 6-month follow-up by at least 10% among smokers with diabetes referred to DEPs compared to standard care.
Time Frame: 26 weeks
Population: One participant from the Intervention (Ottawa Model for Smoking Cessation group) was not included in the analysis as they died during the intervention phase.
Measure: Count of Participants; unit: Participants
Arm/Group | Wait-Listed Control Group | Ottawa Model for Smoking Cessation
Number analyzed (Participants) | 114 | 198
Participants | 3 | 22

2. Secondary Outcome: Cost-effectiveness of Smoking Cessation Interventions.
Description: The cost to implement and maintain the smoking cessation intervention at the patient-level. Cost to implement for patients included program materials, education and counseling.
Time Frame: 26 weeks
Population: The per patient cost was calculated along with the per patient cost for those who did not want to quit smoking.
Measure: Number; unit: Dollars (CAD)
Groups:
- Implementation Cost - Patient: Per-patient cost to implement program
- Implementation Cost - Patient Not Ready to Quit: Per-patient cost for those who are not ready to quit smoking
Arm/Group | Implementation Cost - Patient | Implementation Cost - Patient Not Ready to Quit
Number analyzed (Participants) | 199 | 111
Dollars (CAD) | 262 | 49

3. Other Pre Specified Outcome: Implementation Costs - Clinic
Description: The cost to implement the smoking cessation intervention were calculated a the clinic level. This included all costs related to staff training and program materials.
Time Frame: 26 weeks
Population: The number of clinics included in the analysis
Measure: Number; unit: Dollars (CAD)
Units Other Than Participants: Diabetes Clinics
Groups:
- Implementation Costs - Clinic: The cost to implement and maintain the smoking cessation intervention at the clinic level.
Arm/Group | Implementation Costs - Clinic
Number analyzed (Participants) | NA
Number analyzed (Diabetes Clinics) | 7
Dollars (CAD) | 1870

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from baseline to 6 months.
Description: This was a low risk study. Diabetes clinics were asked to implement a smoking cessation program and offer the related services to their patients. This study assessed the implementation of the program (how successful clinics were in implementing the program and actually getting patients to quit smoking).
Arm/Group | Wait-Listed Control Group | Ottawa Model for Smoking Cessation
All-Cause Mortality (participants affected / at risk) | 0/114 | 0/199
Serious Adverse Events (participants affected / at risk) | 0/114 | 0/199
Other Adverse Events (participants affected / at risk) | 0/114 | 0/199

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No